CLINICAL TRIAL: NCT07119372
Title: A Randomized, Open-label, Comparative Clinical Study of the Efficacy and Safety of BCD-131 and Mircera® in the Treatment of Anemia in Patients With Chronic Kidney Disease on Dialysis
Brief Title: Study of the Efficacy and Safety of BCD-131 and Mircera® in the Treatment of Anemia in Patients With Chronic Kidney Disease on Dialysis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCD-131-3
Record Dates: First submitted 2025-08-07; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Anemia; Chronic Kidney Disease; Chronic Kidney Disease Patients on Hemodialysis; Chronic Kidney Disease 5D
Keywords: Chronic Kidney Disease; CKD; Anemia; Erythropoietin; Darbepoetin; Erythropoiesis-stimulating agent; Dialysis; Hemodialysis; Renal anemia
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-131 (Experimental): BCD-131 (pegdarbepoetin beta)
  Interventions: Biological: BCD-131 (pegdarbepoetin beta)
- Mircera (Active Comparator): Mircera (methoxypolyethylene glycol-epoetin beta)
  Interventions: Biological: Mircera (methoxypolyethylene glycol-epoetin beta)

INTERVENTIONS:
Biological: BCD-131 (pegdarbepoetin beta) — BCD-131 (pegdarbepoetin beta), subcutaneous injection; regimen: once every 4 weeks; therapy duration: 52 weeks
  Arms: BCD-131
Biological: Mircera (methoxypolyethylene glycol-epoetin beta) — Mircera (methoxypolyethylene glycol-epoetin beta), subcutaneous injection; regimen: once every 4 weeks; therapy duration: 52 weeks
  Arms: Mircera

SUMMARY:
BCD-131 is pegylated darbepoetin beta. This clinical study BCD-131-3 is a randomized, open-label, phase III study of the efficacy and safety of BCD-131 and Mircera used for the treatment of anemia in end-stage chronic kidney disease (CKD) patients on dialysis.

DETAILED DESCRIPTION:
This clinical study is based on the hypothesis that BCD-131 is non-inferior to Mircera when used for the treatment of anemia in dialysis patients with end-stage CKD after 32 weeks of therapy.

The study is intended to include subjects with stage 5 CKD, receiving dialysis for at least 90 days before signing the ICF (for patients on hemodialysis - a least 3 times per week and at least 12 hours per week of standard hemodialysis), with established dialysis efficacy, with anemia of renal origin, without other causes for anemia (anemia of chronic disease, vitamin B12 deficiency, folic acid deficiency, iron deficiency, etc.).

This is a study of efficacy of BCD-131 as a maintenance therapy, therefore the population includes patients who have been receiving stable doses of erythropoietins (epoetin alfa, epoetin beta or darbepoetin alfa) for at least 3 months prior to signing the informed consent form (ICF) and throughout the screening period and with target hemoglobin level (100-120 g/L) maintained for at least 2 weeks before the ICF signing and at the screening.

The study includes the following periods:

* Screening period (28 days),
* Main period (32 weeks), consisting of dose titration (weeks 0-12) and maintenance therapy (weeks 13-32) - for the primary efficacy analysis
* Extension period (weeks 33-52) - for long-term safety and efficacy assessment
* Follow-up period (weeks 53-56)

ELIGIBILITY:
Inclusion Criteria:

* The patient signed a written ICF for participation in the study.
* Men and women aged 18 to 75 years inclusive at the time of signing the ICF.
* End stage kidney disease (documented).
* The need for dialysis sessions within at least the last 90 days prior to signing the ICF.
* For patients on hemodialysis - hemodialysis procedures should be at least 3 times a week, for a total duration of at least 12 hours a week.
* Documented use of recombinant erythropoietin (epoetin alfa, epoetin beta or darbepoetin alfa) for at least 90 days prior to signing the ICF.
* The dose of recombinant erythropoietins (epoetin alfa or epoetin beta received 1, 2 or 3 times a week, or darbepoetin alfa received once a week/once every 2 weeks) should be stable for at least 90 days prior to signing the ICF and the entire screening period (documented).
* Target hemoglobin level (100-120 g/L inclusive) based on the results of screening examination (two measurements).
* The efficacy of dialysis established at screening or not more than 14 days before signing the ICF (dialysis dose index (Kt/v) ≥1.2 in patients on long-term hemodialysis, and weekly Kt/v ≥1.7 for patients on peritoneal dialysis).
* Transferrin saturation ≥20%, ferritin level >100 ng/mL at screening.
* Cyancobalamine (vitamin B12) and folic acid levels within the laboratory reference values at screening.
* Willingness of patients of both sexes and their sexual partners of childbearing potential to use methods of contraception in accordance with the protocol, starting from signing the informed consent form, throughout the study and for up to 90 days after receiving the last dose of the drug in the clinical study, as well as to refrain from donation of eggs for female subjects or sperm for male subjects during this period.
* The ability of the patient to comply with the Protocol requirements, in the Investigator's opinion.

Exclusion Criteria:

* Any other diagnosed forms of anemia, except for anemia of renal disease, including anemia in chronic diseases (C-reactive protein level >20 mg/L at screening).
* Diagnosed lupus nephritis or chronic kidney disease due to systemic vasculitis.
* Platelet count <100×109/L based on the results of screening examination.
* A high probability of early withdrawal from the study, in particular a planned (i.e., available information about a planned date and/or a suitable donor) kidney transplant surgery during the estimated period of participation in the study.
* A history of severe allergic reactions (anaphylactic shock or multiple drug allergy) according to the patient, and hypersensitivity to recombinant erythropoietins, polyethylene glycol or any components of the study drugs, or to iron (III) hydroxide sucrose complex.
* Vaccination less than 8 weeks before signing the ICF (according to the patient).
* Diagnosed liver cirrhosis.
* HIV infection.
* ALT, AST >3хULN at screening.
* Decompensated heart disease (NYHA Class IV CHF).
* Resistant hypertension.
* Unstable angina.
* History of acute hemolysis episodes.
* Documented hemoglobinopathy, myelodysplastic syndrome, hematological malignancy, pure red cell aplasia.
* Severe secondary hyperparathyroidism (intact PTH>1000 pg/mL at screening) or biopsy-confirmed bone marrow fibrosis (myelofibrosis).
* Documented episodes of gastrointestinal or other bleeding within less than 90 days prior to signing the ICF.
* Documented history of episodes of thrombosis (acute myocardial infarction, stroke, transient ischemic attacks, deep vein thrombosis, pulmonary thromboembolism within less than 6 months before the signing of the ICF, as well as long-term vascular access thrombosis within 30 days before the signing of the ICF.
* Seizure syndrome, including a history of or epilepsy during the screening period.
* Documented major surgery less than 30 days before signing the ICF.
* Documented blood transfusion within less than 90 days prior to signing the ICF.
* Any acute or chronic infections in the stage of exacerbation, as well as other chronic diseases that at the time of signing the informed consent, may adversely affect the patient's safety while using the study therapy in the opinion of the investigator.
* A history of severe depression, suicidal ideation, or attempted suicide.
* Documented malignancies other than cured basal-cell carcinoma and/or cervical carcinoma in situ with a remission duration of more than 5 years at the time of signing the ICF.
* Known alcohol or drug addiction, or current signs of alcohol/drug addiction, which, according to the investigator, is contraindication for the treatment with the test drug/reference drug or limits the treatment adherence.
* Participation in other clinical studies of medicinal products within less than 90 calendar days prior to signing the informed consent form for participation in this study.
* Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects (%) with the target hemoglobin level (100-120 g/L inclusive) | During the assessment period at Weeks 28-32

SECONDARY OUTCOMES:
Proportion of subjects (%) with the target hemoglobin level (100-120 g/L inclusive) during the last month of therapy | Weeks 48-52
Proportion of subjects (%) with a mean hemoglobin level at the time of assessment within the range of ±10 g/L from baseline | Weeks 28-32
Proportion of subjects (%) with a mean hemoglobin level at the time of assessment within the range of ±10 g/L from baseline | Weeks 48-52
Proportion of subjects (%) who required dose adjustment of the test drug/reference drug during the maintenance therapy stage of the main study period | Weeks 12-32
  In the main study period, a dose adjustment is expected during the first 12 weeks of therapy (titration phase), and a maintenance therapy stage is expected during the subsequent weeks of the main study period.
Proportion of subjects (%) who required dose adjustment of the test drug/reference drug during the extension study period | Weeks 33-52
Proportion of subjects (%) who required blood transfusion during the main study period | Weeks 0-32
Proportion of subjects (%) who required blood transfusion during the entire study | Weeks 0-52
The mean hemoglobin level during the main study period | Weeks 0-32
The mean hemoglobin level during the entire study | Weeks 0-52
Proportion of subjects (%) with hemoglobin values greater than 130 g/L and with values greater than 140 g/L during the main study period | Weeks 0-32
Proportion of subjects (%) with hemoglobin values greater than 130 g/L and with values greater than 140 g/L during the entire study | Weeks 0-52
Proportion of subjects with reported AEs/SAEs, which, according to the investigator, are related to the study drugs | Weeks 0-56
Proportion of subjects in each group who developed CTCAE v. 5.0 grade 3-4 AEs, which, in the investigator's opinion, are related to the use of the study drugs | Weeks 0-56
Proportion of subjects in each group who prematurely withdrew due to AEs/SAEs | Weeks 0-56
Frequency of arterial and venous thrombotic complications (cerebrovascular accident, vascular access thrombosis, etc.) | Weeks 0-56
Frequency of non-fatal myocardial infarction, death from cardiovascular diseases, death from any cause | Weeks 0-56
The Proportion of BAb- and NAb-positive Patients | Weeks 0, 12, 24, 36, and 52
  Blood sampling for immunogenicity assessment (binding antibodies [BAbs] or neutralizing antibodies [NAbs]) will be performed before the first injection (Week 0) and then at Weeks 12, 24, 36, and 52

CONTACTS AND LOCATIONS:
Locations (2):
- Minsk Scientific and Practical Center for Surgery, Transplantology and Hematology, Minsk, Belarus
- B. Braun Avitum Russland Clinics Ltd., Saint Petersburg, Russia